CLINICAL TRIAL: NCT05751525
Title: Impact of Timing of Initiation of Sulphonylurea Therapy on Neurodevelopmental Outcomes in Individuals With Intermediate Developmental Delay, Epilepsy and Neonatal Diabetes (iDEND) Syndrome Due to the V59M Mutation in the KCNJ11 Gene
Brief Title: Impact of Sulphonylureas on Neurodevelopmental Outcomes in KCNJ11-related Intermediate Developmental Delay, Epilepsy and Neonatal Diabetes (iDEND) Syndrome
Acronym: iDEND
Status: Recruiting | Type: Observational
Sponsor: Royal Devon and Exeter NHS Foundation Trust (Other)
Collaborators: University of Chicago (Other); University of Bergen (Other); University of Rome Tor Vergata (Other)
Responsible Party: Sponsor
Other Study IDs: 120925
Record Dates: First submitted 2023-01-25; First posted 2023-03-02 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Neurodevelopmental Disorders; Intellectual Disability; Development Delay; ADHD; Autism Spectrum Disorder; Epilepsy
MeSH Terms: conditions — Neurodevelopmental Disorders; Intellectual Disability; Learning Disabilities; Attention Deficit Disorder with Hyperactivity; Autism Spectrum Disorder; Epilepsy | interventions — Sulfonylurea Compounds

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | US Export: No

GROUPS / COHORTS (2):
- Early SU treatment: Patients with permanent neonatal diabetes (PNDM) due to the V59M mutation in the KCNJ11 gene who commenced sulfonylurea therapy in the first twelve months of life.
  Interventions: Drug: Sulfonylurea
- Late SU treatment: Patients with permanent neonatal diabetes (PNDM) due to the V59M mutation in the KCNJ11 gene who commenced sulfonylurea older than the age of twelve months.
  Interventions: Drug: Sulfonylurea

INTERVENTIONS:
Drug: Sulfonylurea — Glibenlclamide / glyburide

SUMMARY:
The goal of this observational study is to learn about the impact of the diabetes drug glibenclamide (glyburide) on neurodevelopment in individuals with iDEND (developmental delay, epilepsy and neonatal diabetes) due to the V59M mutation in the KCNJ11 gene. The main question it aims to answer is whether initiating sulphonylurea (SU) therapy in the first year of life results in better neurodevelopmental outcomes in affected individuals, in comparison to starting therapy later than 12 months of age.

Participants will undergo a neurodevelopmental assessment comprising parental and teacher completion of standardised questionnaires, and where possible face to face neuropsychological testing.

Researchers will compare the outcomes of these standardised tests in the individuals who started SU therapy <12 months of age in comparison to those who started >12 months of age.

DETAILED DESCRIPTION:
Background:

The role of the KATP channel in the pancreas The KATP channel is made up of 4 pore-forming Kir6.2 subunits (encoded by the KCNJ11 gene) and 4 regulatory SUR1 subunits (encoded by the ABCC8 gene). In the pancreas, the KATP channel plays a central role in glucose-stimulated insulin secretion.

KATP channel mutations cause neonatal diabetes that can be treated with oral sulphonylureas Neonatal diabetes is defined as diabetes occurring in the first 6 months of life; it has an incidence of approximately 1 in 200,000 live births. Neonatal diabetes is due to a monogenic defect, and mutations in the KCNJ11 and ABCC8 genes are the commonest cause. These are important to diagnose as over 90% of patients can switch from insulin treatment to an oral sulphonylurea with a resulting improvement in glycaemic control which is maintained long-term.

Central Nervous System features occur in patients with neonatal diabetes due to KATP mutations.

Around 20% of patients with mutations in the KCNJ11 gene have an overt severe neurological phenotype. This is consistent with the expression of the KATP channel in the brain. There is a phenotype/genotype relationship e.g. most patients with the V59M mutation have the intermediate DEND syndrome (iDEND - Developmental delay, Epilepsy and Neonatal Diabetes), with moderate developmental delay and substantial intellectual disability. DEND syndrome is characterised by severe developmental delay and epilepsy diagnosed within the first 12 months of life. People with iDEND syndrome also show hyperactivity, impulsivity, inattention and impaired visuomotor performance. Autism (comprising impaired language and social interaction and restricted/repetitive behaviours), ADHD and anxiety disorders have been reported in individuals with the V59M mutation. Mouse models with V59M mutations have replicated the hyperactive phenotype seen in humans. These finding suggests a possible role for the KATP channel in neurodevelopment.

Previous research suggests earlier initiation of treatment results in more favourable CNS outcomes After switching from insulin to oral sulphonylureas, some patients with a V59M mutation have a clear but incomplete improvement in neurological / cognitive function suggesting that the KATP channel in the CNS responds in part to sulphonylureas. Sulphonylurea therapy is also associated with changes in brain perfusion patterns, in particular improved cerebellar perfusion. The timing of initiation of sulphonylurea therapy appears to be important; one study showed an inverse correlation between age of initiation of treatment with sulphonylureas and performance in the visual-motor integration test (a neuromotor coordination task) in patients with V59M/A mutations. Another prospective study showed improved neurological and psychomotor function in a group of patients with a mixture of KATP channel mutations (only one of which was V59M); this improvement was greater in the younger patients.

The reason for greater neurological improvements in younger patients may relate to greater neuroplasticity in the brain in the first 12 months of life; if this is the case then it is crucial to make a genetic diagnosis of KATP channel neonatal diabetes early and transfer patients as soon as possible to sulphonylurea therapy.

Despite its clinical importance, to date there has been no formal study of whether age of first treatment with a sulphonylurea affects neurodevelopmental outcomes in patients with V59M mutations.

Aim:

To establish whether early treatment with sulphonylureas improves neurodevelopmental outcomes in patients with the V59M mutation in the KCNJ11 gene.

Objectives:

1. To identify and recruit the largest international cohort of individuals with V59M mutations reported to date.
2. To characterise the neurodevelopmental phenotype in these patients using standardised validated questionnaires and assessments.
3. To compare outcomes in those who started treatment with SU in the first 12 months of life vs those who started treatment later than 12 months.

Methods:

Data collection form will be completed by clinicians / researchers using parent/carer report and / or review of notes +/- clinical observation. The study procedure for each participant is as follows:

* Standard medical, perinatal and social history including major milestones
* Developmental Assessment (see below)

  * Development and Wellbeing Assessment (DAWBA) to establish ICD-10/DSM-IV / V psychiatric diagnoses and Strengths and Difficulties Questionnaire (SDQ) to provide a quantitative measure of psychiatric morbidity in five key areas (hyperactivity, emotional, conduct problems, peer relationships, prosocial behaviour) and overall impact. The DAWBA and SDQ are standardised, validated questionnaires given to informants (usually parents and teachers) and patients themselves if aged 11 years or over and able to complete them. These can be completed online, and normative data derived from large population surveys is available.
  * Leiter-3 International Performance Scale Cognitive battery where neither the examiner nor the child is required to speak, and the child is not required to read or write either. As the test is nonverbal, it is especially suitable for children and adolescents who are cognitively delayed, disadvantaged, nonverbal or non-English speaking, speech or hearing impaired, motor impaired, have a diagnosis of ADHD or autism. Provides IQ scores and scaled scores for its subtests.
  * CCC-2 (Children's Communication Checklist) - parental questionnaire used to identify communication problems in children aged 4-16.

Data analysis:

Patients will be divided into 2 groups based on starting SU treatment (1) >12 months and (2) <12 months. Where possible scores on the above tests will be converted to SD scores using normative population data. Results from the 2 groups will be compared using non-parametric statistical methods to establish whether, for the same mutation, the age at which treatment is initiated impacts on the degree of developmental delay, psychopathology and impact.

ELIGIBILITY:
Inclusion Criteria:

* Current age ≥2 years
* Heterozygous for a V59M mutation in the KCNJ11 gene
* Successfully transferred to oral sulphonylurea therapy
* Willing to participate

Exclusion Criteria:

* Never able to transfer to oral sulphonylurea therapy
* Unwilling to participate

Ages: 2 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Participating centres will recruit and assess participants meeting study eligibility criteria (University of Exeter, UK, University of Chicago, USA, University of Bergen, Norway and University of Rome, Italy). Participants will be allocated to the early treatment or late treatment group depending on age at initiation of SU therapy, in a ratio of 1:2 (early:late).
Sampling Method: Probability Sample
Enrollment: 21 (Estimated)
Dates: Start 2016-07-01 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Number and type of neurodevelopmental and psychiatric disorders | At or up to 2 years after recruitment
  Measured by Development and Wellbeing Assessment (DAWBA)
Level of difficulty due to neurodevelopmental and psychiatric morbidity | At or up to 2 years after recruitment
  Measured by Strengths and Difficulties Questionnaire (SDQ) total difficulties score. Scores range from 0-40 with higher scores indicating greater difficulties. Scores will be converted to Z-scores using normative population data for the purposes of analysis.
Impact on daily life | At or up to 2 years after recruitment
  Measured by SDQ impact score. Scores range from 0-10 for parent and self-report and 0-6 for teacher report, with higher scores indicating greater difficulties. Scores will be converted to Z-scores using normative population data for the purposes of analysis.
IQ score | Up to 3 years after recruitment
  Measured by Leiter-3 International Performance Scale

SECONDARY OUTCOMES:
Major milestones | At or up to 2 years after recruitment
  Measured by parent report / review of clinical records
Communication difficulties | Up to 3 years after recruitment
  Measured by the Children's Communication Checklist 2 (CCC-2) questionnaire, consisting of 70 items scored by parents / caregivers. Lower scores indicate more communication difficulties.
Hyperactivity, emotional problems, conduct problems, peer relationships, prosocial behaviour. | At or up to 2 years after recruitment
  Measured by SDQ subsections. Scores range from 0-10 for each subsection with higher scores indicating greater difficulties, except prosocial score where lower scores indicate greater difficulties. Scores will be converted to Z-scores using normative population data for the purposes of analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Prof Andrew Hattersley, Principal Investigator — University of Exeter / Royal Devon University Healthcare Trust
Locations (4):
- University of Chicago, Chicago, Illinois, United States
- University of Rome, Rome, Italy
- University of Bergen, Bergen, Norway
- University of Exeter, Exeter, United Kingdom

REFERENCES:
- [Background] Gloyn AL, Pearson ER, Antcliff JF, Proks P, Bruining GJ, Slingerland AS, Howard N, Srinivasan S, Silva JM, Molnes J, Edghill EL, Frayling TM, Temple IK, Mackay D, Shield JP, Sumnik Z, van Rhijn A, Wales JK, Clark P, Gorman S, Aisenberg J, Ellard S, Njolstad PR, Ashcroft FM, Hattersley AT. Activating mutations in the gene encoding the ATP-sensitive potassium-channel subunit Kir6.2 and permanent neonatal diabetes. N Engl J Med. 2004 Apr 29;350(18):1838-49. doi: 10.1056/NEJMoa032922. PMID 15115830
- [Background] Pearson ER, Flechtner I, Njolstad PR, Malecki MT, Flanagan SE, Larkin B, Ashcroft FM, Klimes I, Codner E, Iotova V, Slingerland AS, Shield J, Robert JJ, Holst JJ, Clark PM, Ellard S, Sovik O, Polak M, Hattersley AT; Neonatal Diabetes International Collaborative Group. Switching from insulin to oral sulfonylureas in patients with diabetes due to Kir6.2 mutations. N Engl J Med. 2006 Aug 3;355(5):467-77. doi: 10.1056/NEJMoa061759. PMID 16885550
- [Background] Bowman P, Sulen A, Barbetti F, Beltrand J, Svalastoga P, Codner E, Tessmann EH, Juliusson PB, Skrivarhaug T, Pearson ER, Flanagan SE, Babiker T, Thomas NJ, Shepherd MH, Ellard S, Klimes I, Szopa M, Polak M, Iafusco D, Hattersley AT, Njolstad PR; Neonatal Diabetes International Collaborative Group. Effectiveness and safety of long-term treatment with sulfonylureas in patients with neonatal diabetes due to KCNJ11 mutations: an international cohort study. Lancet Diabetes Endocrinol. 2018 Aug;6(8):637-646. doi: 10.1016/S2213-8587(18)30106-2. Epub 2018 Jun 4. PMID 29880308
- [Background] Flanagan SE, Edghill EL, Gloyn AL, Ellard S, Hattersley AT. Mutations in KCNJ11, which encodes Kir6.2, are a common cause of diabetes diagnosed in the first 6 months of life, with the phenotype determined by genotype. Diabetologia. 2006 Jun;49(6):1190-7. doi: 10.1007/s00125-006-0246-z. Epub 2006 Apr 12. PMID 16609879
- [Background] Gloyn AL, Diatloff-Zito C, Edghill EL, Bellanne-Chantelot C, Nivot S, Coutant R, Ellard S, Hattersley AT, Robert JJ. KCNJ11 activating mutations are associated with developmental delay, epilepsy and neonatal diabetes syndrome and other neurological features. Eur J Hum Genet. 2006 Jul;14(7):824-30. doi: 10.1038/sj.ejhg.5201629. Epub 2006 May 3. PMID 16670688
- [Background] Svalastoga P, Sulen A, Fehn JR, Aukland SM, Irgens H, Sirnes E, Fevang SKE, Valen E, Elgen IB, Njolstad PR. Intellectual Disability in KATP Channel Neonatal Diabetes. Diabetes Care. 2020 Mar;43(3):526-533. doi: 10.2337/dc19-1013. Epub 2020 Jan 13. PMID 31932458
- [Background] Bowman P, Broadbridge E, Knight BA, Pettit L, Flanagan SE, Reville M, Tonks J, Shepherd MH, Ford TJ, Hattersley AT. Psychiatric morbidity in children with KCNJ11 neonatal diabetes. Diabet Med. 2016 Oct;33(10):1387-91. doi: 10.1111/dme.13135. Epub 2016 May 21. PMID 27086753
- [Background] Landmeier KA, Lanning M, Carmody D, Greeley SAW, Msall ME. ADHD, learning difficulties and sleep disturbances associated with KCNJ11-related neonatal diabetes. Pediatr Diabetes. 2017 Nov;18(7):518-523. doi: 10.1111/pedi.12428. Epub 2016 Aug 24. PMID 27555491
- [Background] Clark RH, McTaggart JS, Webster R, Mannikko R, Iberl M, Sim XL, Rorsman P, Glitsch M, Beeson D, Ashcroft FM. Muscle dysfunction caused by a KATP channel mutation in neonatal diabetes is neuronal in origin. Science. 2010 Jul 23;329(5990):458-61. doi: 10.1126/science.1186146. Epub 2010 Jul 1. PMID 20595581
- [Background] Mlynarski W, Tarasov AI, Gach A, Girard CA, Pietrzak I, Zubcevic L, Kusmierek J, Klupa T, Malecki MT, Ashcroft FM. Sulfonylurea improves CNS function in a case of intermediate DEND syndrome caused by a mutation in KCNJ11. Nat Clin Pract Neurol. 2007 Nov;3(11):640-5. doi: 10.1038/ncpneuro0640. PMID 17982434
- [Background] Slingerland AS, Nuboer R, Hadders-Algra M, Hattersley AT, Bruining GJ. Improved motor development and good long-term glycaemic control with sulfonylurea treatment in a patient with the syndrome of intermediate developmental delay, early-onset generalised epilepsy and neonatal diabetes associated with the V59M mutation in the KCNJ11 gene. Diabetologia. 2006 Nov;49(11):2559-63. doi: 10.1007/s00125-006-0407-0. Epub 2006 Sep 19. PMID 17047922
- [Background] Slingerland AS, Hurkx W, Noordam K, Flanagan SE, Jukema JW, Meiners LC, Bruining GJ, Hattersley AT, Hadders-Algra M. Sulphonylurea therapy improves cognition in a patient with the V59M KCNJ11 mutation. Diabet Med. 2008 Mar;25(3):277-81. doi: 10.1111/j.1464-5491.2007.02373.x. PMID 18307455
- [Background] Fendler W, Pietrzak I, Brereton MF, Lahmann C, Gadzicki M, Bienkiewicz M, Drozdz I, Borowiec M, Malecki MT, Ashcroft FM, Mlynarski WM. Switching to sulphonylureas in children with iDEND syndrome caused by KCNJ11 mutations results in improved cerebellar perfusion. Diabetes Care. 2013 Aug;36(8):2311-6. doi: 10.2337/dc12-2166. Epub 2013 Mar 5. PMID 23462667
- [Background] Shah RP, Spruyt K, Kragie BC, Greeley SA, Msall ME. Visuomotor performance in KCNJ11-related neonatal diabetes is impaired in children with DEND-associated mutations and may be improved by early treatment with sulfonylureas. Diabetes Care. 2012 Oct;35(10):2086-8. doi: 10.2337/dc11-2225. Epub 2012 Aug 1. PMID 22855734
- [Background] Beltrand J, Elie C, Busiah K, Fournier E, Boddaert N, Bahi-Buisson N, Vera M, Bui-Quoc E, Ingster-Moati I, Berdugo M, Simon A, Gozalo C, Djerada Z, Flechtner I, Treluyer JM, Scharfmann R, Cave H, Vaivre-Douret L, Polak M; GlidKir Study Group. Sulfonylurea Therapy Benefits Neurological and Psychomotor Functions in Patients With Neonatal Diabetes Owing to Potassium Channel Mutations. Diabetes Care. 2015 Nov;38(11):2033-41. doi: 10.2337/dc15-0837. Epub 2015 Oct 5. PMID 26438614